CLINICAL TRIAL: NCT01088997
Title: Milrinone Pharmacokinetics and Pharmacodynamics in Newborns With Persistent Pulmonary Hypertension of the Newborn - a Pilot Study to Enable a Randomized Trial of Intervention
Brief Title: Pharmacokinetic Study of Milrinone in Babies With Persistent Pulmonary Hypertension of the Newborn
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Bedford Pharmaceuticals (Industry); American Medical Association (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-007384
Record Dates: First submitted 2010-03-12; First posted 2010-03-18 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Persistent Fetal Circulation Syndrome
Keywords: Persistent pulmonary hypertension of newborn; PPHN; Persistent pulmonary hypertension; Pulmonary hypertension; Pulmonary hypertension of newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Hypertension, Pulmonary | interventions — Milrinone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Milrinone (Experimental): Subjects will receive a bolus intravenous (IV) infusion of 50 mcg/kg/min of milrinone lactate over 1 hour followed by a continuous IV infusion of 0.5 mcg/kg/min milrinone lactate over 24 hours. After completion of infusion, subjects will be monitored for an additional 24 hours.
  Interventions: Drug: Milrinone Lactate
- Low Dose Milrinone (Experimental): Subjects will receive a bolus intravenous (IV) infusion of 20 mcg/kg/min of milrinone lactate over 1 hour followed by a continuous IV infusion of 0.2 mcg/kg/min milrinone lactate over 24 hours. After completion of infusion, subjects will be monitored for an additional 24 hours.
  Interventions: Drug: Milrinone Lactate

INTERVENTIONS:
Drug: Milrinone Lactate — Milrinone lactate will be given first as an IV bolus over one hour at the assigned dose level, followed by a 24 hour IV infusion at the assigned dose level.
  Other Names: Milrinone

SUMMARY:
The purpose of this pilot study is to determine a safe dose of milrinone to use in a larger study of babies with persistent pulmonary hypertension of the newborn (PPHN).

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn (PPHN) is a condition in which the pulmonary vasculature fails to relax after birth resulting in severe hypoxemia. This condition has a high rate of mortality and morbidity. The current standard of care is treatment with inhaled nitric oxide (iNO). However, for many babies this treatment does not provide sufficient improvement in oxygenation.

In this study, subjects already receiving nitric oxide will be randomized to one of two dosing regimens of milrinone. They will receive milrinone IV for 24 hours and will be monitored for 24 hours afterwards. During this time, milrinone assays will be performed by blood sampling. Echocardiograms will also be performed to explore the pharmacodynamics of milrinone. Safety monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 34 weeks
* Post-natal age < 10 days
* Hypoxemia defined by: Oxygenation Index (OI) >15 (Mean Airway Pressure x Fraction of Inspired Oxygen (FiO2) x 100 /PaO2) as drawn from two post-ductal arterial blood gas samples (in-dwelling arterial catheter) taken at least 15 minutes apart. OR mechanically ventilated and with >75% FiO2 for >6 hours while on iNO
* Absence of congenital heart disease based on a two-dimensional echocardiogram and/or clinical assessment
* An in-dwelling arterial catheter to facilitate painless sampling
* Currently on iNO or plan to start iNO before enrollment

Exclusion Criteria:

* Lethal non-cardiac congenital anomalies including diaphragmatic hernia
* Clinically apparent bleeding; thrombocytopenia <30,000 or other laboratory evidence of coagulopathy
* Currently on extracorporeal membrane oxygenation (ECMO)or plan to initiate ECMO within 2 hours of enrollment

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Michigan/Hutzel Women's Hospital, Detroit, Michigan
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in June 2010 at three large academic medical centers. The study was closed to enrollment at all sites in November 2013.
Groups:
- High Dose Milrinone: Subjects received a 50 mcg/kg loading dose of milrinone lactate given intravenously (IV) over 1 hour followed by an IV infusion of 0.5 mcg/kg/min over 24 hours.
- Low Dose Milrinone: Subjects received a 20 mcg/kg loading dose of milrinone lactate given intravenously (IV) over 1 hour followed by an IV infusion of 0.2 mcg/kg/min over 24 hours.
Period: Overall Study
Arm/Group | High Dose Milrinone | Low Dose Milrinone
Started | 7 | 5
Completed | 4 | 2
Not Completed | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Req. Extracorporeal membrane oxygenation | 1 | 1
Not completed — Excluded prior to receiving drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Dose Milrinone: Subjects received a 50mcg/kg loading dose of milrinone lactate given intravenously (IV) over 1 hour followed by an IV infusion of 0.5mcg/kg over 24 hours
- Low Dose Milrinone: Subjects received a 20mcg/kg loading dose of milrinone lactate given intravenously (IV) over 1 hour followed by an IV infusion of 0.2mcg/kg over 24 hours
- Total: Total of all reporting groups
Arm/Group | High Dose Milrinone | Low Dose Milrinone | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 2 | 4
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Secondary Outcome: Change in Oxygenation Index (OI) From Baseline to up to 24 Hours After Start of Milrinone Infusion
Description: Oxygenation Index (mean airway pressure*Fraction of Inspired Oxygen/Partial Pressure of Oxygen in the blood) was calculated at baseline and every 6 hours after start of infusion until 12-24 hours after initiation of milrinone infusion.
Time Frame: for up to 24 hours after start of infusion
Population: OI was calculated every 6 hours after start of infusion for 24 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Dose Milrinone: 7 subjects were enrolled into this arm, of these only 4 completed study treatment.
- Low Dose Milrinone: 5 subjects were enrolled into this arm, of these only 2 completed study treatment.
Arm/Group | High Dose Milrinone | Low Dose Milrinone
Number analyzed (Participants) | 4 | 2
units on a scale | 4.9 (11.5) | 36.5 (27.0)

2. Primary Outcome: Define Plasma Concentration-time Profile of Milrinone in Neonates With Persistent Pulmonary Hypertension of the Newborn (PPHN) - Clearance (CL, mL/Min)
Description: The schedule of milrinone pharmacokinetic (PK) sampling varied by weight to minimize blood sampling. For babies weighing less than 3kg, samples were drawn at the end of the bolus, 15 minutes prior to the end of infusion (EOI) and 20 minutes, 1, 2, 6 and 12 hours after EOI. For babies weighing 3kg or more, samples were drawn at the end of the bolus, 6 hours after start of infusion, 15 minutes prior to the EOI and 30 minutes, 1, 3, 9 and 15 hours after EOI. Milrinone plasma concentrations were determined using a validated high-performance mass spectrometry assay.
Time Frame: End of bolus dose, 15 minutes prior to end of infusion (EOI), at four time points after EOI with final sample at 12-15 hours after EOI (timing based on infant's weight)
Population: The pharmacokinetic analysis, including the primary outcome parameter, Clearance, was planned a priori to include all the participants pooled together. A PK analysis by arm wouldn't be appropriate. The randomization arms were only created to explore the secondary clinical and pharmacodynamic outcomes.
Measure: Mean (Standard Error); unit: mL/min/3.4 kg
Groups:
- Milrinone Population: Population model developed based on 6 subjects who completed study treatment and were deemed evaluable.
Arm/Group | Milrinone Population
Number analyzed (Participants) | 6
mL/min/3.4 kg | 7.65 (18.8)

3. Secondary Outcome: Change in Myocardial Performance Index (MPI) From Baseline to up to 24 Hours After Start of Milrinone Infusion
Description: An echocardiogram obtained while on milrinone was obtained with the goal of attempting to look for improvements in parameters associated with pulmonary hypertension. The primary parameter measured was the myocardial performance index (MPI). An Echocardiogram was performed at baseline (pre-infusion) and repeated 12-24 hours ater the initiation of the Milrinone infusion. Also known as the Tei index, the MPI is an index that incorporates both systolic and diastolic time intervals in expressing global systolic and diastolic ventricular function. Systolic dysfunction prolongs preejection (isovolumic contraction time, IVCT) and a shortening of the ejection time (ET). Both systolic and diastolic dysfunction result in abnormality in myocardial relaxation which prolongs the relaxation period (isovolumic relaxation time, IVRT). Normal value for MPI is 0.39+/-0.05 with dilated cardiomyopathy value of MPI at 0.59+/-0.10 (both units on a scale)
Time Frame: Up to 24 hours after start of infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Dose Milrinone: 7 subjects were enrolled into the study, of these 4 completed study treatment.
- Low Dose Milrinone: 5 subjects were enrolled into the study, of these 2 completed study treatment and only 1 received 2 MPI measurements
Arm/Group | High Dose Milrinone | Low Dose Milrinone
Number analyzed (Participants) | 4 | 1
units on a scale | -.12 (0.29) | -.09 (0)

ADVERSE EVENTS:
Time Frame: Adverse event assessment was performed continuously from baseline (pre-infusion) through 24 hours after the completion of the milrinone infusion (total of 48 hours).
Description: Included vital signs (i.e., blood pressure, measured hourly per standard of care), cardiorespiratory monitoring (ii.e., cardiac rhythm monitored continuously per standard of care), laboratory data (arterial blood gas collected ever 4 hours; hematology and serum chemistry collected every 24 hours), and head ultrasound (pre/post infusion).
Groups:
- High Dose Milrinone: Subjects received a bolus intravenous (IV) infusion of 50 mcg/kg/min of milrinone lactate over 1 hour followed by a continuous IV infusion of 0.5 mcg/kg/min milrinone lactate over 24 hours.
- Low Dose Milrinone: Subjects received a bolus intravenous (IV) infusion of 20 mcg/kg/min of milrinone lactate over 1 hour followed by a continuous IV infusion of 0.2 mcg/kg/min milrinone lactate over 24 hours.
Arm/Group | High Dose Milrinone | Low Dose Milrinone
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 4/7 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Milrinone (N=7) | Low Dose Milrinone (N=5)
Hypoxia requiring ECMO (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal insufficiency (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Renal and urinary disorders) | 0 | 1
Elevated Liver Function Tests (Hepatobiliary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study enrollment was terminated early resulting in a small number of evaluable subjects for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes